CLINICAL TRIAL: NCT06766175
Title: Impact of Chronic Cough on Activities of Daily Living and Response to Acute High-intensity Exercise
Status: Recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: Hull York Medical School (Unknown); King's College Hospital NHS Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Oliver Price, Associate Professor, University of Leeds
Other Study IDs: 344527
Record Dates: First submitted 2024-12-13; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Chronic Cough (CC)
Keywords: Cough; Physical activity; Exercise; Physiology
MeSH Terms: conditions — Chronic Cough; Cough; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic cough as per European Respiratory Society definition (>8 weeks duration)

SUMMARY:
Chronic cough is a common and debilitating condition that affects up to 10% of the global population. The health impact of chronic cough is multifaceted and manifests both physical and psychological symptoms including syncope, chest pain, lethargy, depression and anxiety. It is now also recognised that chronic cough often leads to social isolation and may impact an individual's ability or confidence to undertake routine daily tasks / lead an active lifestyle.

The primary aim of this study is therefore to characterise the impact of unexplained chronic cough on the ability to undertake daily activities - i.e., determine whether individuals with chronic cough exhibit impaired levels of physical activity during usual daily living when compared with healthy age, gender and BMI matched controls. A secondary aim is to assess the short-term impact of high-intensity exercise on cough (i.e., determine whether an acute bout of exercise alters cough frequency and/or severity).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Chronic cough as per European Respiratory Society definition (>8 weeks duration)
* High symptom burden (i.e., cough visual analogue scale >40 mm at pre-study screening)
* Chest radiograph or CT within 3 years of the screening visit with no abnormalities considered to contribute to chronic cough

Exclusion Criteria:

* Smokers or individuals who gave up smoking within 12 months
* Smoking history >20 pack-years
* Long-COVID or post-COVID syndrome (defined as symptoms lasting over 12-weeks in duration)
* Recent exacerbation of cough within 4 weeks of inclusion
* Respiratory tract infection within 4 weeks of inclusion
* Currently taking any of the following medications:

  * ACE inhibitors and within 3 months of inclusion
  * Antitussives (opioids, pregabalin, gabapentin, amitriptyline, nortriptyline, or over the-counter medications) within 2 weeks of inclusion
  * Medical treatments for gastro-oesophageal reflux disease (GORD), eosinophilic bronchitis or other cough related conditions, initiated or changed (i.e., not in a stable regimen) for 4 weeks prior to inclusion
* Medical history of asthma or exercise-induced bronchoconstriction (EIB), COPD, or chronic bronchitis in the judgement of the investigator
* Medical conditions/history or other circumstances which, in the judgement of the investigators, could increase the risk of adverse events or bias the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with unexplained chronic cough will be recruited from the Hull Cough Clinic, Castle Hill Hospital.
Sampling Method: Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity status assessed using objective wearable accelerometer (ActiGraph LEAP) | 1-week
  Physical activity status including:
  - Absolute daily steps

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No